CLINICAL TRIAL: NCT00209560
Title: A Phase III, Randomized, Open-label Study to Assess the Safety and Efficacy of AQUAVAN® Injection Versus Midazolam HCl for Sedation in Patients Undergoing Minor Surgical Procedures
Brief Title: A Study of AQUAVAN® Injection in the Presence of Pre-Medication in Patients Undergoing Minor Surgical Procedures
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Collaborators: PPD Development, LP (Industry); Covance (Industry)
Responsible Party: Eisai Medical Services, Eisai Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3000-0412
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Results first posted 2012-06-19 (Estimated); Last update posted 2015-01-09 (Estimated); Status verified 2014-07

CONDITIONS: Arthroscopy; Bunionectomy; Osteotomy; Carpal Tunnel
Keywords: AQUAVAN® Injection; Midazolam; Minor surgical procedures; Sedation
MeSH Terms: conditions — Median Neuropathy | interventions — fospropofol

INTERVENTIONS:
Drug: fospropofol disodium

SUMMARY:
The purpose of this study is to determine the safety, tolerability, and efficacy of AQUAVAN® Injection when used for mild-to-moderate sedation in patients undergoing minor surgical procedures.

DETAILED DESCRIPTION:
Randomized, open label, multi-center,midazolam adaptive dose ranging study, in which several dose levels of AQUAVAN® Injection and fentanyl citrate injection will be investigated to produce a desired sedation level in patients undergoing minor surgical and/or therapeutic procedures. A desired sedative dose/dose range and dosing paradigm will be identified based on pre-set criteria using the Modified Observer's Assessment of Alertness/Sedation (OAA/S). The desired sedative dose/dose range and dosing paradigm of AQUAVAN® Injection is defined as one that consistently provides mild to moderate sedation (Modified OAA/S between 2 and 4 inclusive) in majority of patients who are pre-medicated with fentanyl citrate injection.

Midazolam is the most widely used i.v. agent for minimal-to-moderate sedation. The dose range of midazolam to induce minimal to moderate sedation was based on standard clinical practice.

[new paragraph] All patients were pre-medicated with fentanyl citrate as an analgesic.

The outpatient setting has become increasingly popular for various types of medical procedures requiring sedation. In outpatient minor surgical procedures, sedation agents are used to provide mild-to-moderate sedation and are used with other medicines for pain management. Surgeons have searched for alternative treatments to use in the outpatient setting that would provide a faster recovery time with minimal post-procedure amnesia. This injection is used following pretreatment with fentanyl citrate for pain management.

ELIGIBILITY:
Inclusion Criteria:

1. Patient provided signed/dated Informed Consent and HIPAA Authorization after receiving a full explanation of the extent and nature of the study.
2. Patient was at least 18 years of age at the time of screening. (Prior to Amendment 1, dated 03 February 2005, this criterion restricted enrollment to patients who were ≥18 and ≤65 years of age. To ensure that safe dosing levels were administered to patients >65 years of age, AQUAVAN and midazolam dosing levels were reduced when compared with patients between 18 and 65 years of age, inclusive. The majority of patients were enrolled prior to 03 February 2005.)
3. Female patient must have been surgically sterile, postmenopausal, or not pregnant or lactating, and must have been using an acceptable method of birth control for at least 1 month prior to dosing, with a negative urine pregnancy test result at screening and predosing periods.
4. Patient met the American Society of Anesthesiologists (ASA) Physical Status Classification System of I to III.
5. Patient may have been an inpatient or outpatient scheduled to undergo a single minor surgical and/or therapeutic procedure.

Exclusion Criteria:

1. Patient had a history of allergic reaction or hypersensitivity to any anesthetic agent, narcotic, or benzodiazepine.
2. Patient did not meet nils per os (NPO) status per ASA Guideline or institution's guideline.
3. Patient had condition(s) that, in the opinion of the Investigator, could interfere with appropriate airway management.
4. Patient had participated in an investigational drug study within 1 month prior to study start.
5. Patient had a history of mental or visual impairment that would not permit successful measurement of cognitive evaluations.
6. Patient was unwilling to adhere to pre- and postprocedural instructions.
7. The use of fentanyl or midazolam was contraindicated for the patient.
8. Patient had experienced multiple concurrent injuries or trauma.
9. Patient was scheduled to undergo multiple same-day procedures (eg, bunionectomies on both feet).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2004-10; Study Completion 2005-03

CONTACTS AND LOCATIONS:
Overall Officials: James Jones, MD, PharmD, Study Director — Eisai Inc.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study recruited at 18 centers in the US during the period of 29-Oct-2004 to 24 Mar 2005.
Pre-assignment Details: After enrollment and before randomization all subjects, irrespective of treatment group assignment,received fentanyl citrate injection 0.5 µg/kg to 1 µg/kg(based on age)as an analgesic pretreatment 5 minutes prior to the administration of either fospropofol disodium (Also known as,LUSEDRA and formerly known as AQUAVAN) or midazolam midazolam HCl).
Groups:
- Fospropofol Disodium: 525 mg to 980 mg (dose based on weight and age): one initial intravenous (i.v.) bolus dose. Supplemental doses of fospropofol disodium 105 mg to 140 mg (based on weight and age) were administered as needed.
- Midazolam: 0.5 to 2 mg (dose based on weight and age): one initial i.v. bolus dose. Supplemental doses of midazolam 0.25 mg to 1 mg (based on weight and age) were administered as needed.
Period: Overall Study
Arm/Group | Fospropofol Disodium | Midazolam
Started | 121 | 42
Completed | 120 | 42
Not Completed | 1 | 0
Not completed — Lack of Efficacy | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fospropofol Disodium | Midazolam | Total
Number analyzed (Participants) | 121 | 42 | 163
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.3 (11.0) | 45.3 (11.5) | 45.3 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84 | 24 | 108
  Male | 37 | 18 | 55
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 14 | 3 | 17
  Other | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 19 | 10 | 29
  White | 87 | 28 | 115
  More than one race | 0 | 0 | 0
Weight (kg) [Number; unit: particpants]
  <55 | 7 | 0 | 7
  55 to > 80 | 41 | 14 | 55
  >80 | 73 | 28 | 101
American Society of Anesthesiologists Status (ASA) [Number; unit: particpants]
  I (A normal healthy patient) | 48 | 19 | 67
  II (A patient with mild systemic disease) | 71 | 21 | 92
  III (A patient with severe systemic disease) | 2 | 2 | 4
History of Adverse Reactions following a Previous Sedation [Number; unit: participants]
  Yes | 3 | 2 | 5
  No | 111 | 37 | 148
  No history of sedation | 7 | 3 | 10

OUTCOME MEASURES:

1. Primary Outcome: Successful Sedation of Subjects, Defined for a Subject as Having 3 Consecutive Scores ≤ 4 on the Modified Observer's Assessment of Alertness/Sedation Scale and Completing the Procedure w/o Alternative Sedative Medications/w/o Manual/Mechanical Ventilation
Description: The Modified OAA/S (MOAA/S) scale is based on a validated, 6-point rating scale. Scores are not combined.
  Score 5 (alert) -- responds readily to name spoken in normal tone Score 4 -- Lethargic response to name spoken in normal tone Score 3 -- Responds only after name is called loudly and/or repeatedly Score 2 -- Responds only after mild prodding or shaking Score 1 -- Responds only after painful trapezius squeeze Score 0 -- Does not respond to painful trapezius squeeze
Time Frame: Sedation success was assessed at 2 minute intervals until the end of the procedure
Population: The pP1 and mITT population included all subjects randomized,received either fospropofol disodium or midazolam, had at least 1 postdose clinical assessment, and were not terminated due to the Investigator's decision for nonstudy drug related findings. A 95% confidence interval for the sedation success rate was calculated for each treatment group.
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Fospropofol Disodium | Midazolam
Number analyzed (Participants) | 121 | 42
participants
  pPI Population Sedation Success | 94.2 (94.2) [88.4 to 97.6] | 78.6 [63.2 to 89.7]
  mITT Population Sedation Success | 94.2 [88.4 to 97.6] | 78.6 [63.2 to 89.7]

2. Secondary Outcome: Time to Fully Alert From the End of the Procedure
Description: Time to Fully Alert, defined as the time to the first of 3 consecutive Modified OAA/S scores of 5 from the end of the surgical procedure, was summarized.
Time Frame: At 2-minute intervals from the end of the procedure until the subject met the criteria for Fully Alert status
Population: The primary analysis for the secondary efficacy endpoint was based on the mITT population. Missing values or incomplete data were not imputed.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Fospropofol Disodium | Midazolam
Number analyzed (Participants) | 120 | 42
minutes | 8.4 (10.9) | 4.1 (5.4)

ADVERSE EVENTS:
Arm/Group | Fospropofol Disodium | Midazolam
Serious Adverse Events (participants affected / at risk) | 1/121 | 0/42
Other Adverse Events (participants affected / at risk) | 104/121 | 31/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fospropofol Disodium (N=121) | Midazolam (N=42)
Appendictis (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fospropofol Disodium (N=121) | Midazolam (N=42)
Anal discomfort (Gastrointestinal disorders) | 3 | 0
Constipation (Gastrointestinal disorders) | 5 | 2
Nausea (Gastrointestinal disorders) | 19 | 7
Pruritus ani (Gastrointestinal disorders) | 3 | 0
Vomiting (Gastrointestinal disorders) | 7 | 3
Chills (General disorders) | 2 | 0
Pain (General disorders) | 6 | 3
Incision site complication (Injury, poisoning and procedural complications) | 5 | 6
Post procedural pain (Injury, poisoning and procedural complications) | 63 | 18
Procedural complication (Injury, poisoning and procedural complications) | 12 | 3
Alanine aminotransfersase increased (Investigations) | 4 | 0
Aspartate aminotransferase increased (Investigations) | 3 | 0
Gamma-glutamyltransferase increased (Investigations) | 3 | 0
Hepatic enzyme increased (General disorders) | 5 | 0
White blood cell count increased (General disorders) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 | 5
Burning sensation (Nervous system disorders) | 2 | 0
Dizziness (Nervous system disorders) | 4 | 0
Dysgeusia (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 6 | 0
Paraesthesia (Nervous system disorders) | 19 | 1
Genital burning sensation (Reproductive system and breast disorders) | 7 | 0
Paraesthesia of genital female (Reproductive system and breast disorders) | 2 | 0
Pruritus genital (Reproductive system and breast disorders) | 5 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 23 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 21 | 0
Pruritus generalized (Skin and subcutaneous tissue disorders) | 5 | 0
Hypotension (Vascular disorders) | 4 | 0

LIMITATIONS AND CAVEATS:
Analysis of results from a previous fospropofol study (3000-0410) completed during the enrollment of this study indicated that the dosing regimen needed to be re-evaluated. The study was prematurely terminated after 168 subjects were randomized.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No